CLINICAL TRIAL: NCT05968183
Title: The Value of HPV Testing for Cervical Cancer Screening in Women Living With HIV
Brief Title: The Value of HPV Testing for Cervical Cancer Screening in Women Living With HIV (PAPILLO-VIH)
Acronym: PAPILLO-VIH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: CHSD_0026_MATER; 2022-A01844-39 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-07-04; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: HIV Seropositivity
Keywords: HPV test; cervical cancer
MeSH Terms: conditions — HIV Seropositivity; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to evaluate the interest of a screening strategy based on the HPV test in patients living with HIV, compared to the cell smear alone in the same population.

The Secondary objective of this study is to verify if the use of HPV testing could allow for a longer follow-up of these patients in case of negativity, and thus allow for a standardization of clinicians' practices.

DETAILED DESCRIPTION:
Since 2019, a new screening strategy has been implemented and is based on high-risk, HPV tests, which, when negative, allow for spaced monitoring in the general population after age 30 (every 5 years instead of every 3 years.)

These tests therefore allow for earlier detection of patients at risk but also for longer follow-up when they are negative.

To our knowledge, there is currently no evaluation of HPV testing as part of routine screening in patients living with HIV.

The recommendations for this population are based on the use of the cervico-vaginal smear with cytological analysis. The smear should be taken every year and surveillance may be repeated every 3 years. If there are 3 consecutive smears without abnormalities and a controlled viral load with CD4 counts > 500 mm3. In practice, many patients do not meet these criteria and must, therefore, undergo annual screening; the increase in the number of smears also leads to an increase in the number of second-line examinations such as colposcopy.

Since there is no recommendation for HPV testing in this population, the use of dual detection (cytology and HPV testing) is left to the discretion of the clinician.

By mutual agreement with the clinicians of the maternity department of the Saint-Denis Hospital (CHSD), this double detection was introduced in 2021, using the same sample (single swab for both analyses: cytology and HPV test).

Therefore, it seems interesting to verify the possibility of a screening strategy based on HPV testing in patients living with HIV, by correlating the results of HPV testing and cell smears in the population of patients living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Women living with HIV
* Age 25-65 years
* Managed in the CHSD maternity ward: consultation or hospitalization
* Having signed a consent form

Exclusion Criteria:

* Age ≤ 24 years, or ≥ 66 years
* Women who are not HIV positive
* Patients under legal protection (guardianship, curatorship)
* Patients deprived of liberty
* Patients not affiliated to a social security system
* Refusal to participate in the research

Ages: 25 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Cohort of patients who have been living with HIV seen in maternity consultations
  over 1 year at our institution.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Demographic characteristics | Day 1
HIV history | Day 1
medical history | Day 1
comorbidities | Day 1
clinical examination data | Day 1

SECONDARY OUTCOMES:
Results of HPV Cytology | Day 1
Results of cell smear | Day 1
Results of additional examinations prescribed | Day 1
  Results of any additional examinations prescribed

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Denis, Saint-Denis, France

REFERENCES:
- [Background] Laara E, Day NE, Hakama M. Trends in mortality from cervical cancer in the Nordic countries: association with organised screening programmes. Lancet. 1987 May 30;1(8544):1247-9. doi: 10.1016/s0140-6736(87)92695-x. PMID 2884378
- [Background] Koliopoulos G, Nyaga VN, Santesso N, Bryant A, Martin-Hirsch PP, Mustafa RA, Schunemann H, Paraskevaidis E, Arbyn M. Cytology versus HPV testing for cervical cancer screening in the general population. Cochrane Database Syst Rev. 2017 Aug 10;8(8):CD008587. doi: 10.1002/14651858.CD008587.pub2. PMID 28796882
- [Background] Srisomboon S, Tantipalakorn C, Muangmool T, Srisomboon J. Risk of High-Grade Cervical Lesions in Atypical Squamous Cells of Undetermined Significance (ASC-US) Cytology: Comparison between HIV-Infected and HIV-Negative Women. Asian Pac J Cancer Prev. 2021 Feb 1;22(2):547-551. doi: 10.31557/APJCP.2021.22.2.547. PMID 33639672
- [Background] Denslow SA, Rositch AF, Firnhaber C, Ting J, Smith JS. Incidence and progression of cervical lesions in women with HIV: a systematic global review. Int J STD AIDS. 2014 Mar;25(3):163-77. doi: 10.1177/0956462413491735. Epub 2013 Aug 29. PMID 24216030
- [Background] Liu G, Sharma M, Tan N, Barnabas RV. HIV-positive women have higher risk of human papilloma virus infection, precancerous lesions, and cervical cancer. AIDS. 2018 Mar 27;32(6):795-808. doi: 10.1097/QAD.0000000000001765. PMID 29369827
- [Background] Sakdadech N, Muangmool T, Srisomboon J. HIV-Infected Women with Low-Grade Squamous Intraepithelial Lesion on Cervical Cytology Have Higher Risk of Underlying High-Grade Cervical Intraepithelial Neoplasia. Int J Environ Res Public Health. 2021 Sep 28;18(19):10211. doi: 10.3390/ijerph181910211. PMID 34639509
- [Background] Nappi L, Carriero C, Bettocchi S, Herrero J, Vimercati A, Putignano G. Cervical squamous intraepithelial lesions of low-grade in HIV-infected women: recurrence, persistence, and progression, in treated and untreated women. Eur J Obstet Gynecol Reprod Biol. 2005 Aug 1;121(2):226-32. doi: 10.1016/j.ejogrb.2004.12.003. Epub 2005 Jan 18. PMID 16054967
- [Background] Gupta K, Philipose CS, Rai S, Ramapuram J, Kaur G, Kini H, Gv C, Adiga D. A Study of Pap Smears in HIV-Positive and HIV-Negative Women from a Tertiary Care Center in South India. Acta Cytol. 2019;63(1):50-55. doi: 10.1159/000496211. Epub 2019 Feb 5. PMID 30721904
- [Background] Hawes SE, Critchlow CW, Sow PS, Toure P, N'Doye I, Diop A, Kuypers JM, Kasse AA, Kiviat NB. Incident high-grade squamous intraepithelial lesions in Senegalese women with and without human immunodeficiency virus type 1 (HIV-1) and HIV-2. J Natl Cancer Inst. 2006 Jan 18;98(2):100-9. doi: 10.1093/jnci/djj010. PMID 16418512
- [Background] Keller MJ, Burk RD, Xie X, Anastos K, Massad LS, Minkoff H, Xue X, D'Souza G, Watts DH, Levine AM, Castle PE, Colie C, Palefsky JM, Strickler HD. Risk of cervical precancer and cancer among HIV-infected women with normal cervical cytology and no evidence of oncogenic HPV infection. JAMA. 2012 Jul 25;308(4):362-9. doi: 10.1001/jama.2012.5664. PMID 22820789
- [Background] Clifford GM, Goncalves MA, Franceschi S; HPV and HIV Study Group. Human papillomavirus types among women infected with HIV: a meta-analysis. AIDS. 2006 Nov 28;20(18):2337-44. doi: 10.1097/01.aids.0000253361.63578.14. PMID 17117020
- [Background] Harris TG, Burk RD, Palefsky JM, Massad LS, Bang JY, Anastos K, Minkoff H, Hall CB, Bacon MC, Levine AM, Watts DH, Silverberg MJ, Xue X, Melnick SL, Strickler HD. Incidence of cervical squamous intraepithelial lesions associated with HIV serostatus, CD4 cell counts, and human papillomavirus test results. JAMA. 2005 Mar 23;293(12):1471-6. doi: 10.1001/jama.293.12.1471. PMID 15784870